CLINICAL TRIAL: NCT00747487
Title: A Double-Blind, Randomised, Placebo-Controlled Study of the Efficacy, Safety and Tolerability of Idebenone in the Treatment of Patients With Leber's Hereditary Optic Neuropathy
Brief Title: Study to Assess Efficacy,Safety and Tolerability of Idebenone in the Treatment of Leber's Hereditary Optic Neuropathy
Acronym: RHODOS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Santhera Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SNT-II-003
Record Dates: First submitted 2008-09-04; First posted 2008-09-05 (Estimated); Last update posted 2013-05-27 (Estimated); Status verified 2013-05

CONDITIONS: Leber's Hereditary Optic Neuropathy
Keywords: Leber; LHON; Leber's Hereditary Optic Neuropathy; Idebenone
MeSH Terms: conditions — Optic Atrophy, Hereditary, Leber | interventions — idebenone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Idebenone
  Interventions: Drug: Idebenone
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Idebenone — Idebenone 900 mg/day
  Arms: 1
Drug: Placebo — Placebo
  Arms: 2

SUMMARY:
This study is meant to assess the effectiveness of idebenone on visual function measures in patients with Leber's Hereditary Optic Neuropathy over a 6 months period.

DETAILED DESCRIPTION:
The study involves 6 clinic visits.

ELIGIBILITY:
Inclusion Criteria:

* Age > or = 14 years and < 65 years
* Impaired visual acuity in at least one eye due to LHON
* Onset of visual loss due to LHON lies five years or less prior to Baseline
* Confirmation of either G11778A, T14484C or G3460A LHON mtDNA mutations at >60% in blood
* No explanation for the visual failure besides LHON
* Body weight ≥ 45 kg
* Negative urine pregnancy test at Screening and at Baseline (women of childbearing potential).

Exclusion Criteria:

* Treatment with Coenzyme Q10 or idebenone within 1 month prior to Baseline
* Pregnancy and/or breast-feeding
* Weekly alcohol intake 35 units (men) or 24 units (women)
* Current drug abuse
* Clinically significant abnormalities of clinical haematology or biochemistry including, but not limited to, elevations greater than 2 times the upper limit of normal of AST, ALT or creatinine
* Participation in another clinical trial of any investigational drug within 3 months prior to Baseline
* Other factor that, in the investigator's opinion, excludes the patient from entering the study

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2007-11; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Best recovery of logMAR visual acuity between baseline and Week 24 in either right or left eye | 24 weeks

SECONDARY OUTCOMES:
Change in the patient's best logMAR visual acuity between baseline and week 24 | 24 weeks
Change in scotoma area in both eyes | Day -1, Week 4, Week 12, Week 24
Change in optic nerve fibre layer thickness in both eyes | Day -1, Week 4, Week 12, Week 24
Colour contrast sensitivity in both eyes (in a subset of patients) | Day -1, Week 4, Week 12, Week 24
logMAR visual acuity as a continuous variable in both eyes | Screening, Day -1, Week 4, Week 12, Week 24, Week 28
Clinical Global Impression of Change | Week 4, Week 12 and Week 24
Change in Health-Related Quality of Life (HRQOL) | Day -1, Week 4, Week 12, Week 24
Change in self-reported general energy levels | Day -1, Week 4, Week 12, Week 24, Week 28
Proportion of patients in which visual acuity in the initially least affected eye does not deteriorate to 1.0 log MAR or more ( in LHON patients with eye still less affected than 0.5 logMAR at trial entry) | 24 weeks
Plasma levels of idebenone matched to measures of efficacy and safety | 24 weeks
• Best visual acuity at Week 24 (best eye at Week 24) compared to best visual acuity at Baseline (best eye at Baseline) | 24 weeks
• Count of eyes/ patients for which the visual acuity improves between baseline and week 24 | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Prof Patrick F Chinnery, MD, Principal Investigator — Clinical Research Facility, 4th Floor Leazes Wing, Royal Victoria Infirmary; Prof Thomas Klopstock, MD, Principal Investigator — Klinikum der Universität München - Grosshadern, Neurologische Klinik und Poliklinik
Locations (3):
- Unité de recherche clinique Ophtalmologie- Hopital Notre-Dame, Montreal, Quebec, Canada
- Klinikum der Universität München - Grosshadern, Neurologische Klinik und Poliklinik, Munich, Germany
- Clinical Research Facility, 4th Floor Leazes Wing, Royal Victoria Infirmary, Newcastle upon Tyne, United Kingdom

REFERENCES:
- [Result] Klopstock T, Yu-Wai-Man P, Dimitriadis K, Rouleau J, Heck S, Bailie M, Atawan A, Chattopadhyay S, Schubert M, Garip A, Kernt M, Petraki D, Rummey C, Leinonen M, Metz G, Griffiths PG, Meier T, Chinnery PF. A randomized placebo-controlled trial of idebenone in Leber's hereditary optic neuropathy. Brain. 2011 Sep;134(Pt 9):2677-86. doi: 10.1093/brain/awr170. Epub 2011 Jul 25. PMID 21788663
- [Result] Rudolph G, Dimitriadis K, Buchner B, Heck S, Al-Tamami J, Seidensticker F, Rummey C, Leinonen M, Meier T, Klopstock T. Effects of idebenone on color vision in patients with leber hereditary optic neuropathy. J Neuroophthalmol. 2013 Mar;33(1):30-6. doi: 10.1097/WNO.0b013e318272c643. PMID 23263355
- See also: Website for LHON patients in Canada — http://www.santhera.com/index.php?mid=101&vid=&lang=en
- See also: Website for LHON patients in Germany — http://www.nefo.med.uni-muenchen.de/Forschungshauptseite/klinstudien/therapeutic-trial-of-idebenone-in-lhon